CLINICAL TRIAL: NCT04431453
Title: A Phase 2/3 Single-Arm, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Remdesivir (GS-5734™) in Participants From Birth to < 18 Years of Age With COVID-19
Brief Title: Study of Remdesivir in Participants Below 18 Years Old With COVID-19
Acronym: CARAVAN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-540-5823; 2020-001803-17 (EudraCT Number)
Expanded Access: NCT04323761 (Approved for marketing)
Record Dates: First submitted 2020-06-08; First posted 2020-06-16 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg (Experimental): Participants will receive RDV 200 mg, intravenous (IV) infusion on Day 1 followed by RDV 100 mg, IV infusion, daily, up to 10 days.
  Interventions: Drug: Remdesivir
- RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg (Experimental): Participants will receive RDV 5 mg/kg, IV infusion on Day 1 followed by RDV 2.5 mg/kg mg, IV infusion, daily, up to 10 days.
  Interventions: Drug: Remdesivir
- RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg (Experimental): Participants will receive RDV 5 mg/kg, IV infusion on Day 1 followed by RDV 2.5 mg/kg mg, IV infusion, daily, up to 10 days.
  Interventions: Drug: Remdesivir
- RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg (Experimental): Participants will receive RDV 5 mg/kg, IV infusion on Day 1 followed by RDV 2.5 mg/kg mg, IV infusion, daily, up to 10 days.
  Interventions: Drug: Remdesivir
- RDV, Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg (Experimental): Participants will receive RDV 5 mg/kg, IV infusion on Day 1 followed by RDV 2.5 mg/kg mg, IV infusion, daily, up to 10 days.
  Interventions: Drug: Remdesivir
- RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg (Experimental): Participants will receive RDV 2.5 mg/kg, IV infusion on Day 1 followed by RDV 1.25 mg/kg mg, IV, daily, up to 10 days.
  Interventions: Drug: Remdesivir
- RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg (Experimental): Participants will receive RDV 2.5 mg/kg, IV infusion on Day 1 followed by RDV 1.25 mg/kg mg, IV, daily, up to 10 days.
  Interventions: Drug: Remdesivir
- RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg (Experimental): Participants will receive RDV 200 mg, IV infusion on Day 1 followed by RDV 100 mg, IV infusion daily up to 10 days.
  Interventions: Drug: Remdesivir

INTERVENTIONS:
Drug: Remdesivir — Administered as an intravenous infusion
  Other Names: GS-5734™; Veklury®

SUMMARY:
The goals of this clinical study are to learn more about the study drug, remdesivir, and how safe it is in participants less than 18 years old with coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
Pediatric participants will be enrolled as follows:

Pediatric participants ≥ 28 days to < 18 years old:

* Cohort 1: ≥ 12 years to < 18 years and weight ≥ 40 kg
* Cohort 2: ≥ 28 days to < 18 years and weight ≥ 20 kg to < 40 kg
* Cohort 3: ≥ 28 days to < 18 years and weight ≥ 12 kg to < 20 kg
* Cohort 4: ≥ 28 days to < 18 years and weight ≥ 3 kg to < 12 kg
* Cohort 8: < 12 years and weight ≥ 40 kg

Term neonatal participants 0 days to < 28 days old:

* Cohort 5: ≥ 14 days to < 28 days of age, gestational age > 37 weeks and weight at screening ≥ 2.5 kg
* Cohort 6: 0 days to < 14 days of age, gestational age > 37 weeks and birth weight ≥ 2.5 kg

Preterm neonates and infants 0 days to < 56 days old:

* Cohort 7: 0 days to < 56 days of age, gestational age ≤ 37 weeks and birth weight ≥ 1.5 kg

ELIGIBILITY:
Key Inclusion Criteria:

* Aged < 18 years of age who meet one of the following weight criteria (where permitted according to local law and approved nationally and by relevant institutional review board (IRB) or independent ethics committee (IEC)).

  * a) Cohort 1: ≥ 12 years to < 18 years of age and weight at screening ≥ 40 kg
  * b) Cohorts 2-4: ≥ 28 days to < 18 years of age and weight at screening ≥ 3 kg and < 40 kg
  * c) Cohort 5: ≥ 14 days to < 28 days of age, gestational age > 37 weeks and weight at screening ≥ 2.5 kg
  * d) Cohort 6: 0 days to < 14 days of age, gestational age > 37 weeks and birth weight of ≥ 2.5 kg
  * e) Cohort 7: 0 days to < 56 days of age, gestational age ≤ 37 weeks and birth weight of ≥ 1.5 kg
  * f) Cohort 8: < 12 years of age and weight at screening ≥ 40 kg
* Severe acute respiratory syndrome coronavirus (SARS-CoV-2) infection confirmed by polymerase chain reaction (PCR).
* Hospitalized and requiring medical care for coronavirus disease 2019 (COVID-19).

Key Exclusion Criteria:

* Concurrent treatment with other agents with actual or possible direct antiviral activity against SARS-CoV-2 < 24 hours prior to study drug dosing.
* Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 X upper limit of normal (ULN).
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m^2 using Schwartz formula for individuals ≥ 1 year of age.
* Creatinine above protocol specified thresholds for < 1 year of age.
* Positive pregnancy test at Screening only for female of child bearing potential. Note: If female participants who become pregnant during the study or are discovered to be pregnant after receiving at least one dose may continue study drug, after discussion with the investigator.
* On renal replacement therapies (intermittent hemodialysis (iHD), peritoneal dialysis (PD), continuous renal replacement therapy (CRRT)).

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (32):
- United States (22):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Ronald Reagan University of California, Los Angeles Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UC Davis Medical center, Sacramento, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Tampa General Hospital (Inpatient Visits), Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Spectrum Health/Helen De Vos Children's Hospital, Grand Rapids, Michigan
  - Children's Minnesota, Minneapolis, Minnesota
  - Northwell Health-Cohen Children's Medical Center, New Hyde Park, New York
  - NYC Health + Hospitals/Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center-Levine Children's Hospital, Charlotte, North Carolina
  - Lehigh Valley Hospital/Lehigh Valley Health Network (LVH/LVHN), Allentown, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
- Italy (3):
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - Azienda Ospedaliera di Padova - Dipartimento Salute della Donna e del Bambino, Padua
  - UO Clinica Pediatrica, Ospedale Pietro Barilla - AOU di Parma, Parma
- Spain (6):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
- Alder Hey Children's NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Background] Ahmed A, Rojo P, Agwu A, Kimberlin D, Deville J, Mendez-Echevarria A, et al. Remdesivir Treatment for COVID-19 in Hospitalized Children: CARAVAN Interim Results [Presentation]. European Congress of Clinical Microbiology & Infectious Diseases (ECCMID) 2022; 2022 23-26 April; Lisbon, Portugal and Online.
- [Background] Ahmed A, Rojo P, Agwu A, Kimberlin D, Deville J, Mendez-Echevarria A, et al. Remdesivir Treatment for COVID-19 in Hospitalized Children: CARAVAN Interim Results [Presentation]. Virtual Conference on Retroviruses and Opportunistic Infections (CROI) 2022; 2022c 12-16 February.
- [Background] Munoz F, Muller W, Ahmed A, Kimberlin D, Mendez-Echevarria A, Chen JS, et al. Safety and efficacy of Remdesivir in a pediatric COVID-19 population (CROI) [Abstract 617]. Topics in antiviral medicine 2021;29 (1):237.
- [Background] Pikora C, Bamford A, Luzuriaga K, Wiznia A, Rojo Conejo P, Muller B, et al. Challenges of remdesivir pediatric development for SARS-CoV-2 infection in a pandemic. 12th International Workshop on HIV Pediatrics; 2020 November 16-17; Virtual Event.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-540-5823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Italy, Spain, the United Kingdom, and the United States.
Pre-assignment Details: 60 participants were screened.
Groups:
- Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg: Participants received RDV 200 mg, intravenous (IV) infusion on Day 1 followed by RDV 100 mg, IV infusion daily up to 10 days.
- RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg; RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg; RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg; RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg: Participants received RDV 5 mg/kg, IV infusion on Day 1 followed by RDV 2.5 mg/kg mg, IV infusion daily up to 10 days.
- RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg; RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg: Participants received RDV 2.5 mg/kg, IV infusion on Day 1 followed by RDV 1.25 mg/kg mg, IV infusion daily up to 10 days.
- RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg: Participants received RDV 200 mg, IV infusion on Day 1 followed by RDV 100 mg, IV infusion daily up to 10 days.
Period: Overall Study
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Started | 12 | 12 | 12 | 12 | 4 | 1 | 1 | 5
Completed | 11 | 11 | 11 | 9 | 3 | 1 | 1 | 4
Not Completed | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 1
Not completed — Withdrew Consent | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Enrolled but Never Treated | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug.
Groups:
- Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg: Participants received RDV 200 mg, intravenous (IV) infusion on Day 1 followed by RDV 100 mg, IV infusion, daily, up to 10 days.
- RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg; RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg; RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg; RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg: Participants received RDV 5 mg/kg, IV infusion on Day 1 followed by RDV 2.5 mg/kg mg, IV infusion, daily, up to 10 days.
- RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg; RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg: Participants received RDV 2.5 mg/kg, IV infusion on Day 1 followed by RDV 1.25 mg/kg mg, IV infusion, daily, up to 10 days.
- RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg: Participants received RDV 200 mg, IV infusion on Day 1 followed by RDV 100 mg, IV infusion, daily, up to 10 days.
- Total: Total of all reporting groups
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 1 | 1 | 5 | 58
Age, Customized [Count of Participants; unit: Participants] — Population: Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
  Participants
    number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    Newborns (0-27 days) | 0 | 0 | 0 | 0 | 3 |  |  | 0 | 3
    Infants and toddlers (28 days-23 months) | 0 | 0 | 1 | 12 | 0 |  |  | 0 | 13
    Children (2-11 years) | 0 | 8 | 11 | 0 | 0 |  |  | 5 | 24
    Adolescents (12-17 years) | 12 | 4 | 0 | 0 | 0 |  |  | 0 | 16
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
  Participants
    number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    Female | 8 | 7 | 5 | 7 | 1 |  |  | 3 | 31
    Male | 4 | 5 | 7 | 5 | 2 |  |  | 2 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
  Participants
    number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    Hispanic or Latino | 3 | 7 | 7 | 3 | 0 |  |  | 3 | 23
    Not Hispanic or Latino | 8 | 5 | 5 | 9 | 3 |  |  | 2 | 32
    Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 |  |  | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
  Participants
    number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0
    Black or African American | 5 | 2 | 4 | 2 | 0 |  |  | 1 | 14
    White | 7 | 9 | 6 | 8 | 3 |  |  | 3 | 36
    More than one race | 0 | 1 | 2 | 2 | 0 |  |  | 1 | 6
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
  participants
    United States: number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    United States | 9 | 11 | 9 | 9 | 2 |  |  | 3 | 43
    United Kingdom: number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    United Kingdom | 0 | 0 | 0 | 1 | 0 |  |  | 0 | 1
    Italy: number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    Italy | 0 | 0 | 0 | 1 | 1 |  |  | 1 | 3
    Spain: number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    Spain | 3 | 1 | 3 | 1 | 0 |  |  | 1 | 9
Number of Participants With Clinical Status (7-Point Ordinal Scale) Score [Count of Participants; unit: Participants] — The 7-point ordinal scale is an assessment of the clinical status of participant at a given study day:1. Death;2.Hospitalized,on invasive mechanical ventilation or extracorporeal membrane oxygenation(ECMO);3.Hospitalized, on noninvasive ventilation or high-flow oxygen devices;4.Hospitalized,requiring low-flow supplemental oxygen;5.Hospitalized,not requiring supplemental oxygen - requiring ongoing medical care(COVID-19 related or otherwise);6.Hospitalized,not requiring supplemental oxygen - no longer requiring ongoing medical care(other than per-protocol RDV administration);7.Not hospitalized. Population: Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
  Participants
    number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    Score 1 | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0
    Score 2 | 1 | 3 | 3 | 5 | 2 |  |  | 0 | 14
    Score 3 | 6 | 4 | 3 | 3 | 1 |  |  | 2 | 19
    Score 4 | 2 | 3 | 0 | 3 | 0 |  |  | 2 | 10
    Score 5 | 3 | 2 | 6 | 0 | 0 |  |  | 1 | 12
    Score 6 | 0 | 0 | 0 | 1 | 0 |  |  | 0 | 1
    Score 7 | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0
Oxygen Support Status [Count of Participants; unit: Participants] — Oxygen support status was derived from the 7-point ordinal scale, 1 = death; 2 = invasive mechanical ventilation; 3 = high flow oxygen; 4 = low flow oxygen; 5 or 6 = room air; 7 = discharge. Participants with Baseline oxygen status for scores: 2 'invasive mechanical ventilation'; 3 'High Flow Oxygen'; 4 'Low Flow Oxygen', and 5 or 6 'Room Air' are reported. Population: Participants with oxygen support status were analyzed. Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
  Participants
    number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    High Flow Oxygen | 6 | 4 | 3 | 3 | 1 |  |  | 2 | 19
    Low Flow Oxygen | 2 | 3 | 0 | 3 | 0 |  |  | 2 | 10
    Room Air | 3 | 2 | 6 | 1 | 0 |  |  | 1 | 13
    Invasive Mechanical Ventilation Status | 1 | 3 | 3 | 5 | 2 |  |  | 0 | 14
Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) Ribonucleic Acid (RNA) Viral Load [Mean (Standard Deviation); unit: log10 copies per mL] — The assessment were done for the samples: nasal/oropharyngeal (OP), nasopharyngeal (NP)/oropharyngeal (OP), endotracheal (ET) tube aspirates, and rectal/fecal swabs. Population: Participants with data available for the specific category were analyzed. Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
  log10 copies per mL
    Nasal/oropharyngeal Swabs: number analyzed (Participants) | 5 | 5 | 4 | 3 | 1 | 0 | 0 | 1 | 19
    Nasal/oropharyngeal Swabs | 5.35 (1.796) | 4.87 (2.807) | 3.18 (0.967) | 5.41 (2.165) | 5.02 (NA) — SD cannot be calculated for 1 participant. |  |  | 6.20 (NA) — SD cannot be calculated for 1 participant. | 4.80 (1.998)
    Nasopharyngeal/oropharyngeal Swabs: number analyzed (Participants) | 5 | 4 | 5 | 7 | 2 | 0 | 0 | 4 | 27
    Nasopharyngeal/oropharyngeal Swabs | 5.93 (2.172) | 5.37 (1.879) | 5.67 (2.273) | 5.55 (1.854) | 5.99 (0.183) |  |  | 6.12 (1.628) | 5.78 (1.802)
    Endotracheal Tube Aspirates: number analyzed (Participants) | 1 | 4 | 2 | 3 | 1 | 0 | 0 | 0 | 11
    Endotracheal Tube Aspirates | 5.36 (NA) — SD cannot be calculated for 1 participant. | 5.58 (3.554) | 6.09 (0.840) | 6.68 (1.540) | 4.63 (NA) — SD cannot be calculated for 1 participant. |  |  |  | 5.87 (2.180)
    Rectal/fecal Swabs: number analyzed (Participants) | 8 | 7 | 8 | 11 | 3 | 0 | 0 | 5 | 42
    Rectal/fecal Swabs | 3.30 (1.593) | 2.63 (0.757) | 2.72 (1.034) | 3.84 (1.341) | 4.27 (1.107) |  |  | 2.75 (1.274) | 3.26 (1.297)
Pediatric Early Warning Score (PEWS) Scale Score [Count of Participants; unit: Participants] — Behavior:0=playing;appropriate;1=sleeping;2=irritable;3=lethargic;confused;reduced response to pain. Cardiovascular:0=normal;pink;capillary refill(cr)1-2 seconds(secs);1=Tachycardia< 20 above normal for age;2=Tachycardia 20-29 above normal for age;gray;cr=4 secs;3=Tachycardia >=30 above/bradycardia >=10 below normal for age;Gray;cr>=5 secs.Respiratory:0=Normal;1=Respiratory rate(rr)>10 above normal using accessory muscles;30+%fraction of inspired oxygen(FiO2)/3+L/min;2= rr>20 above normal and retractions;40%FiO2 or 6+L/min;3 =rr>=5 below normal with retractions and grunting;50%FiO2/8+L/min. Population: Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
  Participants
    Behavior: number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    Behavior: Score: 0 | 7 | 6 | 5 | 2 | 0 |  |  | 2 | 22
    Behavior: Score: 1 | 3 | 3 | 2 | 3 | 1 |  |  | 1 | 13
    Behavior: Score: 2 | 1 | 0 | 2 | 3 | 0 |  |  | 1 | 7
    Behavior: Score: 3 | 1 | 3 | 3 | 4 | 2 |  |  | 1 | 14
    Cardiovascular: number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    Cardiovascular: Score: 0 | 9 | 7 | 7 | 8 | 1 |  |  | 2 | 34
    Cardiovascular: Score: 1 | 1 | 2 | 3 | 1 | 2 |  |  | 3 | 12
    Cardiovascular: Score: 2 | 2 | 1 | 0 | 1 | 0 |  |  | 0 | 4
    Cardiovascular: Score: 3 | 0 | 2 | 2 | 2 | 0 |  |  | 0 | 6
    Respiratory: number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5 | 56
    Respiratory: Score: 0 | 4 | 1 | 6 | 4 | 0 |  |  | 2 | 17
    Respiratory: Score: 1 | 2 | 5 | 2 | 0 | 1 |  |  | 0 | 10
    Respiratory: Score: 2 | 3 | 2 | 2 | 3 | 0 |  |  | 1 | 11
    Respiratory: Score: 3 | 3 | 4 | 2 | 5 | 2 |  |  | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug and/or any AEs leading to premature discontinuation of study drug.
Time Frame: From first dose date (Day 1) up to follow-up assessment (maximum duration: 30 days)
Population: Safety Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug.
  Data for Cohorts 6 and 7 were not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5
percentage of participants | 91.7 | 58.3 | 75.0 | 58.3 | 66.7 |  |  | 80.0

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Graded Laboratory Abnormalities
Description: Treatment-emergent graded laboratory abnormalities were defined as values that increase at least 1 toxicity grade from baseline at any time post baseline up to and including the date of last dose of study drug plus 30 days. The laboratory abnormalities were graded using division of allergy and infectious diseases (DAIDS) scale. DAIDS scale is used to grade the severity of adult and pediatric unwanted medical events. Grade 1: mild event, Grade 2: moderate event, Grade: serious event, Grade 4: potentially life-threatening event.
Time Frame: From first dose date (Day 1) up to follow-up assessment (maximum duration: 30 days)
Population: Participants in the Safety Analysis Set with at least 1 postbaseline value for the test under evaluation were analyzed. Data for Cohorts 6 and 7 were not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Number; unit: percentage of participants
Groups:
- Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg; RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg: Participants received RDV 200 mg, IV infusion on Day 1 followed by RDV 100 mg, IV infusion daily up to 10 days.
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 3 | 0 | 0 | 5
percentage of participants
  Any grade | 100 | 83.3 | 91.7 | 90.9 | 100 |  |  | 80
  Grade 3 or 4 | 75 | 16.7 | 41.7 | 36.4 | 100 |  |  | 60

3. Primary Outcome: Pharmacokinetic (PK) Parameter: Cmax of Remdesivir and Its Metabolites GS-704277 and GS-441524 at Steady State
Description: Cmax is defined as maximum plasma concentration of drug. Plasma concentrations were drawn as follows: (1) for Cohorts 1-4 and 8 on Day 2 and Day 3 with Day 5 as optional; (2) for Cohorts 5-7 on Day 2 or Day 3.
Time Frame: Day 2: end of infusion and 4 hours post end of infusion, Day 3: pre-infusion and 2 hours post end of infusion, and Day 5: middle of infusion and 6 hours post end of infusion; infusion duration: 30 minutes to 2 hours
Population: The RDV and Metabolites PK Analysis Set included all enrolled participants who received at least 1 dose of RDV and for whom PK concentrations of RDV and metabolites were available.
  Data for Cohorts 6 and 7 were not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 11 | 10 | 3 | 0 | 0 | 5
ng/mL
  Remdesivir | 4108.7 (1365.15) | 6003.5 (1879.86) | 5980.1 (2284.08) | 5192.9 (2066.65) | 4829.0 (956.16) |  |  | 4235.7 (1790.53)
  GS-704277 | 360.6 (208.11) | 469.0 (239.72) | 484.8 (244.07) | 407.8 (132.45) | 466.0 (110.87) |  |  | 297.9 (160.18)
  GS-441524 | 276.4 (327.14) | 210.5 (121.02) | 186.5 (103.09) | 209.8 (49.73) | 371.8 (151.10) |  |  | 230.4 (255.03)

4. Primary Outcome: PK Parameter: AUCtau of Remdesivir and Its Metabolites GS-704277 and GS-441524 at Steady State
Description: AUCtau is defined as area under the concentration versus time curve over the dosing interval. Plasma concentrations were drawn as follows: (1) for Cohorts 1-4 and 8 on Day 2 and Day 3 with Day 5 as optional; (2) for Cohorts 5-7 on Day 2 or Day 3.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 11 | 10 | 3 | 0 | 0 | 5
h*ng/mL
  Remdesivir | 2630.1 (923.85) | 3937.9 (1981.40) | 6752.1 (10911.98) | 3625.7 (3361.19) | 2650.3 (587.77) |  |  | 2519.6 (1235.49)
  GS-704277 | 1222.9 (1348.12) | 860.3 (512.58) | 876.0 (720.39) | 776.0 (485.18) | 1049.0 (253.73) |  |  | 671.4 (553.30)
  GS-441524 | 5486.2 (7599.27) | 3016.1 (2425.78) | 2751.8 (1868.93) | 2969.1 (940.73) | 6899.3 (3910.28) |  |  | 4336.8 (5692.30)

5. Secondary Outcome: Percentage of Participants With Clinical Improvement on a 7-point Ordinal Scale Score
Description: Clinical improvement was defined as ≥ 1-point and ≥ 2-point improvement from Baseline clinical status or recovery or discharged alive on 7-point ordinal scale. Recovery was defined as an improvement from a Baseline score of 2 - 5 to a score of 6 or 7 or an improvement from a Baseline score of 6 to 7 on the ordinal scale. The ordinal scale was used for the assessment of the clinical status at a given day using a 7-point ordinal scale with an increasing score indicating improvement. Scale: 1=Death, 2=Hospitalized, on invasive mechanical ventilation or ECMO, 3=Hospitalized, on non-invasive ventilation or high flow oxygen devices, 4=Hospitalized, requiring low flow supplemental oxygen, 5=Hospitalized, not requiring supplemental oxygen-requiring ongoing medical care COVID-19 related or otherwise), 6=Hospitalized, not requiring supplemental oxygen-no longer required ongoing medical care (other than RDV administration), 7=Not hospitalized. The 95% CI was based on the Clopper-Pearson method.
Time Frame: Day 10
Population: The Full Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug.
  Data for Cohorts 6 and 7 were not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5
percentage of participants
  ≥ 1-point Improvement from Baseline | 50.0 [21.1 to 78.9] | 91.7 [61.5 to 99.8] | 100.0 [73.5 to 100.0] | 58.3 [27.7 to 84.8] | 33.3 [0.8 to 90.6] |  |  | 80.0 [28.4 to 99.5]
  ≥ 2-point Improvement from Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11 | 3 | 0 | 0 | 5
  ≥ 2-point Improvement from Baseline | 41.7 [15.2 to 72.3] | 91.7 [61.5 to 99.8] | 100.0 [73.5 to 100.0] | 54.5 [23.4 to 83.3] | 33.3 [0.8 to 90.6] |  |  | 80.0 [28.4 to 99.5]
  Recovery | 25.0 [5.5 to 57.2] | 75.0 [42.8 to 94.5] | 91.7 [61.5 to 99.8] | 41.7 [15.2 to 72.3] | 33.3 [0.8 to 90.6] |  |  | 80.0 [28.4 to 99.5]

6. Secondary Outcome: Time (Days) to Discharge From Hospital
Description: Time to discharge was the duration from the first dose date to getting discharged from the hospital.
Time Frame: From first dose date (Day 1) up to follow-up assessment (maximum duration: 30 days)
Population: The participants in the Full Analysis Set who were discharged alive on or prior to Day 30 were analyzed.
  Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg: Participants received RDV 200 mg, intravenous (IV) infusion on Day 1 followed by RDV 100 mg, IV infusion daily up to 10 days.
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5
days | 12 [8 to 24] | 7 [5 to 9] | 5 [4 to 9] | 7 [4 to 19] | NA [9 to NA] — Median and upper bound of range (Q3) could not be calculated because less than 50% and 75% of participants, respectively, experienced the event. Hence the days were reported as NA. |  |  | 10 [4 to 18]

7. Secondary Outcome: Number of Participants With Change From Baseline in Oxygenation Use
Description: Oxygen support status was derived from the 7-point ordinal scale score, 1 = death; 2 = invasive mechanical ventilation; 3 = high flow oxygen; 4 = low flow oxygen; 5 or 6 = room air; 7 = discharge. Change from Baseline for participants with oxygenation use status as '3=High Flow Oxygen', '4=Low Flow Oxygen' and '5=Room Air' at Baseline.
Time Frame: Day 10
Population: Participants in Full Analysis Set with Oxygenation use status as 'High Flow Oxygen', 'Low Flow Oxygen' and 'Room Air' at Baseline were analyzed. Number analyzed are participants applicable for the specific categories.
  Data for Cohorts 6 and 7 were not reported due to participants' confidentiality reasons as there were only 1 participant in each of these groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 11 | 9 | 9 | 7 | 1 | 0 | 0 | 5
Participants
  High flow oxygen (Baseline): number analyzed (Participants) | 6 | 4 | 3 | 3 | 1 | 0 | 0 | 2
  High flow oxygen (Baseline): Death (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0
  High flow oxygen (Baseline): IMV (Day 10) | 2 | 0 | 0 | 0 | 0 |  |  | 1
  High flow oxygen (Baseline): High Flow oxygen (Day 10) | 1 | 0 | 0 | 0 | 0 |  |  | 0
  High flow oxygen (Baseline): Low Flow oxygen (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0
  High flow oxygen (Baseline): Room Air (Day 10) | 2 | 0 | 0 | 0 | 0 |  |  | 0
  High flow oxygen (Baseline): Discharge (Day 10) | 1 | 4 | 3 | 2 | 1 |  |  | 1
  High flow oxygen (Baseline): Missing (Day 10) | 0 | 0 | 0 | 1 | 0 |  |  | 0
  Low Flow Oxygen (Baseline): number analyzed (Participants) | 2 | 3 | 0 | 3 | 0 | 0 | 0 | 2
  Low Flow Oxygen (Baseline): Death (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Low Flow Oxygen (Baseline): IMV (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Low Flow Oxygen (Baseline): High Flow oxygen (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Low Flow Oxygen (Baseline): Low Flow oxygen (Day 10) | 0 | 0 | 0 | 1 | 0 |  |  | 0
  Low Flow Oxygen (Baseline): Room Air (Day 10) | 1 | 0 | 0 | 0 | 0 |  |  | 1
  Low Flow Oxygen (Baseline): Discharge (Day 10) | 1 | 3 | 0 | 2 | 0 |  |  | 1
  Low Flow Oxygen (Baseline): Missing (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Room Air (Baseline): number analyzed (Participants) | 3 | 2 | 6 | 1 | 0 | 0 | 0 | 1
  Room Air (Baseline): Death (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Room Air (Baseline): IMV (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Room Air (Baseline): High Flow oxygen (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Room Air (Baseline): Low Flow oxygen (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Room Air (Baseline): Room Air (Day 10) | 2 | 0 | 0 | 0 | 0 |  |  | 0
  Room Air (Baseline): Discharge (Day 10) | 1 | 2 | 6 | 1 | 0 |  |  | 1
  Room Air (Baseline): Missing (Day 10) | 0 | 0 | 0 | 0 | 0 |  |  | 0

8. Secondary Outcome: Number of Participants With Change From Baseline in the Use of Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO)
Description: Mechanical ventilation status was derived from the 7-point ordinal scale score, 1 = death; 2 = invasive mechanical ventilation; 3 = high flow oxygen; 4 = low flow oxygen; 5 or 6 = room air; 7 = discharge.
Time Frame: Day 10
Population: Participants in Full Analysis Set with Oxygenation use status as 'Mechanical Ventilation or ECMO' at Baseline were analyzed.
  Data for Cohorts 6 and 7 were not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 1 | 3 | 3 | 5 | 2 | 0 | 0 | 0
Participants
  Death | 0 | 0 | 0 | 0 | 0 |  |  |
  Invasive Mechanical ventilation | 1 | 1 | 0 | 2 | 2 |  |  |
  High Flow Oxygen | 0 | 0 | 0 | 0 | 0 |  |  |
  Low Flow Oxygen | 0 | 1 | 0 | 0 | 0 |  |  |
  Room Air | 0 | 0 | 1 | 2 | 0 |  |  |
  Discharge | 0 | 0 | 2 | 0 | 0 |  |  |
  Missing | 0 | 1 | 0 | 1 | 0 |  |  |

9. Secondary Outcome: Days to First Confirmed Negative Polymerase Chain Reaction (PCR) Result
Description: Confirmed negative PCR is defined by as 2 consecutive negative PCR results or negative result at the last available sample for participants who completed or discontinued from the study. The assessment were done for the samples: nasal/oropharyngeal (OP), nasopharyngeal (NP)/oropharyngeal (OP), endotracheal (ET) aspirates, and rectal/fecal swabs.
Time Frame: From first dose date (Day 1) up to follow-up assessment (maximum duration: 30 days)
Population: The Full Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug.
  Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5
days
  Nasal/OP Samples: number analyzed (Participants) | 6 | 5 | 4 | 3 | 1 | 0 | 0 | 5
  Nasal/OP Samples | NA [5 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | 5 [3 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | 7 [5 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | NA [4 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | 10 [10 to 10] |  |  | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA.
  NP/OP Samples: number analyzed (Participants) | 3 | 7 | 7 | 7 | 2 | 0 | 0 | 4
  NP/OP Samples | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | NA [7 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | NA [5 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | NA [10 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. |  |  | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA.
  ET aspirates: number analyzed (Participants) | 2 | 3 | 1 | 3 | 2 | 0 | 0 | 0
  ET aspirates | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | NA [3 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | NA [3 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. |  |  |
  Rectal/Faecal samples: number analyzed (Participants) | 9 | 12 | 11 | 10 | 3 | 0 | 0 | 5
  Rectal/Faecal samples | 5 [3 to 10] | 3 [3 to 5] | 5 [3 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | 7 [5 to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days were reported as NA. | 3 [3 to 5] |  |  | 4 [3 to 7]

10. Secondary Outcome: Change From Baseline in Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) Viral Load Up to Day 10 or Up to the First Confirmed Negative PCR Result
Description: Change from baseline in SARS-CoV-2 viral load up to Day 10 or up to the first negative PCR result with confirmation (whichever comes first) were reported. The assessment were done for the samples: nasal/oropharyngeal (OP) samples, nasopharyngeal (NP)/OP samples, endotracheal (ET) aspirates, and rectal/fecal swabs.
Time Frame: Baseline, Day 10, and Day of Discharge (Day 10 or before)
Population: The Full Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug. Number analyzed are participants with data available for analysis for the specific category.
  Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Mean (Standard Deviation); unit: log10 copies per mL
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5
log10 copies per mL
  Nasal/OP Samples, Change at Day 10: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  Nasal/OP Samples, Change at Day 10 | -3.01 (NA) — SD could not be estimated for 1 participant. |  | 0 (0) |  | -2.36 (NA) — SD could not be estimated for 1 participant. |  |  | -1.76 (NA) — SD could not be estimated for 1 participant.
  Nasal/OP Samples, Change at Discharge: number analyzed (Participants) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
  Nasal/OP Samples, Change at Discharge |  | -4.65 (NA) — SD could not be estimated for 1 participant. |  | -1.56 (1.228) |  |  |  |
  NP/OP Samples, Change at Day 10: number analyzed (Participants) | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 1
  NP/OP Samples, Change at Day 10 |  | -2.17 (2.197) |  | -2.60 (1.283) | -3.28 (0.183) |  |  | 0.46 (NA) — SD could not be estimated for 1 participant.
  NP/OP Samples, Change at Discharge: number analyzed (Participants) | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 3
  NP/OP Samples, Change at Discharge | -2.86 (NA) — SD could not be estimated for 1 participant. | -3.72 (NA) — SD could not be estimated for 1 participant. | -0.87 (1.391) | 1.42 (NA) — SD could not be estimated for 1 participant. |  |  |  | -0.05 (1.184)
  ET aspirates, Change at Day 10: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  ET aspirates, Change at Day 10 |  | -5.94 (NA) — SD could not be estimated for 1 participant. |  |  | -1.92 (NA) — SD could not be estimated for 1 participant. |  |  |
  ET aspirates, Change at Discharge: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rectal or Fecal Swabs, Change at Day 10: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Rectal or Fecal Swabs, Change at Day 10 | 0.38 (NA) — SD could not be estimated for 1 participant. | -0.39 (NA) — SD could not be estimated for 1 participant. |  | -1.87 (NA) — SD could not be estimated for 1 participant. |  |  |  | 1.38 (NA) — SD could not be estimated for 1 participant.
  Rectal or Fecal Swabs, Change at Discharge: number analyzed (Participants) | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 2
  Rectal or Fecal Swabs, Change at Discharge |  | 1.12 (NA) — SD could not be estimated for 1 participant. | -0.09 (1.999) | -1.47 (0.479) |  |  |  | 0 (0)

11. Secondary Outcome: Bilirubin Concentrations in < 14-day-old Participants
Time Frame: From first dose date (Day 1) up to follow-up assessment (maximum duration: 30 days)
Population: Data for Cohorts 6 and 7 were not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Arm/Group | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants With Clinical Improvement Based on Scoring Using the Pediatric Early Warning Score (PEWS) Improvement Scale
Description: The PEWS was measured by 3 components, where 1= behavior, 2= perfusion assessed by capillary refill and heart rate, and 3= respiratory status assessed by respiratory rate, effort, and oxygen requirement. The score ranged between 0 to 9 point, with higher score representing the highest severity level. A negative change from baseline value indicated an improvement. Data are reported for participants with a PEWS behavior score ≥ 2 at baseline, and a ≥ 2-point improvement (indicated by a decrease) in PEWS behavior score by Day 10, participants with a PEWS behavior score ≥ 1 at baseline, with ≥ 1-point improvement in PEWS behavior score by Day 10 and participants who recovered in PEWS behavior, defined as a Baseline score of 1 through 3 improved to a score of 0.
Time Frame: Day 10
Population: The Full Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug. Number analyzed are participants with data available for analysis for the specific category.
  Data for Cohorts 6 and 7 were not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5
percentage of participants
  ≥ 2-point Improvement from Baseline- Respiratory: number analyzed (Participants) | 6 | 6 | 4 | 8 | 2 | 0 | 0 | 3
  ≥ 2-point Improvement from Baseline- Respiratory | 33.3 [4.3 to 77.7] | 83.3 [35.9 to 99.6] | 75.0 [19.4 to 99.4] | 42.9 [9.9 to 81.6] | 0 [0 to 84.2] |  |  | 66.7 [9.4 to 99.2]
  ≥ 1-point Improvement from Baseline- Respiratory: number analyzed (Participants) | 8 | 11 | 6 | 8 | 3 | 0 | 0 | 3
  ≥ 1-point Improvement from Baseline- Respiratory | 50.0 [15.7 to 84.3] | 81.8 [48.2 to 97.7] | 83.3 [35.9 to 99.6] | 42.9 [9.9 to 81.6] | 33.3 [0.8 to 90.6] |  |  | 66.7 [9.4 to 99.2]
  Recovery- Respiratory: number analyzed (Participants) | 8 | 11 | 6 | 8 | 3 | 0 | 0 | 3
  Recovery- Respiratory | 37.5 [8.5 to 75.5] | 81.8 [48.2 to 97.7] | 83.3 [35.9 to 99.6] | 42.9 [9.9 to 81.6] | 33.3 [0.8 to 90.6] |  |  | 66.7 [9.4 to 99.2]
  ≥ 2-point Improvement from Baseline- Behavior: number analyzed (Participants) | 2 | 3 | 5 | 7 | 2 | 0 | 0 | 2
  ≥ 2-point Improvement from Baseline- Behavior | 0 [0 to 84.2] | 33.3 [0.8 to 90.6] | 100 [47.8 to 100] | 66.7 [22.3 to 95.7] | 0 [0 to 84.2] |  |  | 50 [1.3 to 98.7]
  ≥ 1-point Improvement from Baseline- Behavior: number analyzed (Participants) | 5 | 6 | 7 | 10 | 3 | 0 | 0 | 3
  ≥ 1-point Improvement from Baseline- Behavior | 40 [5.3 to 85.3] | 66.7 [22.3 to 95.7] | 100 [59 to 100] | 66.7 [29.9 to 92.5] | 66.7 [9.4 to 99.2] |  |  | 33.3 [0.8 to 90.6]
  Recovery- Behavior: number analyzed (Participants) | 5 | 6 | 7 | 10 | 3 | 0 | 0 | 3
  Recovery- Behavior | 40 [5.3 to 85.3] | 66.7 [22.3 to 95.7] | 100 [59 to 100] | 55.6 [21.2 to 86.3] | 33.3 [0.8 to 90.6] |  |  | 33 [0.8 to 90.6]
  ≥ 2-point Improvement from Baseline- Cardiovascular: number analyzed (Participants) | 2 | 3 | 2 | 3 | 0 | 0 | 0 | 0
  ≥ 2-point Improvement from Baseline- Cardiovascular | 0 [0 to 84.2] | 66.7 [9.4 to 99.2] | 100 [15.8 to 100] | 100 [15.8 to 100] |  |  |  |
  ≥ 1-point Improvement from Baseline- Cardiovascular: number analyzed (Participants) | 3 | 5 | 5 | 4 | 2 | 0 | 0 | 3
  ≥ 1-point Improvement from Baseline- Cardiovascular | 33.3 [0.8 to 90.6] | 80 [28.4 to 99.5] | 100 [47.8 to 100] | 66.7 [9.4 to 99.2] | 50 [1.3 to 98.7] |  |  | 66.7 [9.4 to 99.2]
  Recovery- Cardiovascular: number analyzed (Participants) | 3 | 5 | 5 | 4 | 2 | 0 | 0 | 3
  Recovery- Cardiovascular | 0 [0 to 70.8] | 80 [28.4 to 99.5] | 100 [47.8 to 100] | 33.3 [0.8 to 90.6] | 50 [1.3 to 98.7] |  |  | 66.7 [9.4 to 99.2]

13. Secondary Outcome: Plasma Concentrations of Sulfobutylether β-cyclodextrin Sodium (SBECD)
Description: Plasma concentrations were drawn as follows: (1) for Cohorts 1-4 and 8 on Day 2 and Day 3, with Day 5 as optional; (2) for Cohorts 5-7 on Day 2 or Day 3.
Time Frame: as for outcome 3
Population: The SBECD PK Analysis Set included all participants who were enrolled and received at least 1 dose of RDV and for whom PK concentrations of SBECD were available.
  Data for Cohorts 6 and 7 were not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 11 | 10 | 3 | 0 | 0 | 5
ug/mL
  Day 2, End of Infusion: number analyzed (Participants) | 10 | 12 | 10 | 9 | 1 | 0 | 0 | 5
  Day 2, End of Infusion | 217.7 (262.32) | 173.0 (119.06) | 187.8 (75.89) | 138.3 (104.06) | NA (NA) — Data were not available as the concentrations were below the level of quantification (BLQ). |  |  | 156.6 (57.21)
  Day 2, 4 hours post infusion: number analyzed (Participants) | 10 | 11 | 10 | 9 | 1 | 0 | 0 | 4
  Day 2, 4 hours post infusion | 110.1 (270.72) | 24.3 (23.90) | 14.2 (15.03) | 36.2 (32.75) | NA (NA) — Data were not available as the concentrations were below the level of quantification (BLQ). |  |  | 16.2 (8.31)
  Day 3, Pre-Infusion: number analyzed (Participants) | 10 | 10 | 10 | 8 | 2 | 0 | 0 | 5
  Day 3, Pre-Infusion | 78.5 (209.65) | NA (NA) — Data were not available as the concentrations were below the level of quantification (BLQ). | NA (NA) — Data were not available as the concentrations were below the level of quantification (BLQ). | NA (NA) — Data were not available as the concentrations were below the level of quantification (BLQ). | NA (NA) — Data were not available as the concentrations were below the level of quantification (BLQ). |  |  | NA (NA) — Data were not available as the concentrations were below the level of quantification (BLQ).
  Day 3, 2 hours post infusion: number analyzed (Participants) | 11 | 12 | 9 | 7 | 2 | 0 | 0 | 5
  Day 3, 2 hours post infusion | 90.1 (221.54) | 47.5 (52.62) | 47.4 (38.99) | 58.2 (25.89) | 61.0 (79.20) |  |  | 48.0 (50.41)
  Day 5, Middle of Infusion: number analyzed (Participants) | 6 | 5 | 3 | 5 | 0 | 0 | 0 | 3
  Day 5, Middle of Infusion | 229.0 (221.14) | 105.5 (72.05) | 156.3 (23.12) | 118.2 (121.22) |  |  |  | 184.2 (131.82)
  Day 5, 6 Hours post infusion: number analyzed (Participants) | 3 | 4 | 2 | 4 | 0 | 0 | 0 | 2
  Day 5, 6 Hours post infusion | 141.2 (261.96) | 6.6 (3.15) | NA (NA) — Data were not available as the concentrations were below the level of quantification (BLQ). | 12.4 (9.89) |  |  |  | NA (NA) — Data were not available as the concentrations were below the level of quantification (BLQ).

14. Secondary Outcome: Percentage of Participants With Concomitant Use of Medications Other Than RDV for Treatment of COVID-19
Description: Participants who received at least one concomitant non-study COVID-19 medication from the first day of RDV treatment through the 30-day Follow-up visit or early withdrawal are reported.
Time Frame: first dose date (Day 1) up to follow-up assessment (maximum duration: 30 days)
Population: The Safety Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug.
  Data for Cohorts 6 and 7 were not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 3 | 0 | 0 | 5
percentage of participants | 100.0 | 100.0 | 83.3 | 83.3 | 66.7 |  |  | 100.0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: First dose date up to approximately 8 weeks Adverse events: From first dose date (Day 1) up to follow-up assessment (maximum duration: 30 days)
Description: All-cause mortality: All Enrolled Analysis Set will include all participants who are enrolled into the study.
  Adverse events: Safety Analysis Set included all enrolled participants who received at least one dose of study drug. Data for Cohorts 6 and 7 are not reported due to participants' confidentiality reasons as there was only 1 participant in each of these groups.
Arm/Group | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg. | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg
All-Cause Mortality (participants affected / at risk) | 2/12 | 1/12 | 0/12 | 0/12 | 0/4 | 0/0 | 0/0 | 1/5
Serious Adverse Events (participants affected / at risk) | 5/12 | 2/12 | 0/12 | 3/12 | 1/3 | 0/0 | 0/0 | 1/5
Other Adverse Events (participants affected / at risk) | 11/12 | 7/12 | 9/12 | 7/12 | 2/3 | 0/0 | 0/0 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg (N=12) | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg (N=12) | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg (N=12) | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg. (N=12) | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg (N=3) | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg (N=0) | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg (N=0) | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg (N=5)
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Negative pressure pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemodynamic instability (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remdesivir (RDV), Cohort 1: Age 12 to <18 Years and Weight ≥40 kg (N=12) | RDV, Cohort 2: Age ≥ 28 Days to < 18 Years and Weight ≥ 20 kg to < 40 kg (N=12) | RDV, Cohort 3: Age ≥ 28 Days to < 18 Years and Weight ≥ 12 kg to < 20 kg (N=12) | RDV, Cohort 4: Age ≥ 28 Days to < 18 Years and Weight ≥ 3 kg to < 12 kg. (N=12) | RDV,Cohort 5: Age ≥14 - <28 Days of Age, Gestational Age >37 Weeks, and Weight at Baseline ≥2.5 kg (N=3) | RDV, Cohort 6: Age 0 to < 14 Days of Age, Gestational Age > 37 Weeks, and Birth Weight ≥ 2.5 kg (N=0) | RDV, Cohort 7: Age 0 to < 56 Days of Age, Gestational Age ≤ 37 Weeks, and Birth Weight ≥ 1.5 kg (N=0) | RDV, Cohort 8: < 12 Years and Weight ≥ 40 kg (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery dilatation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Physical deconditioning (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Calcium ionised decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin C decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device leakage (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT04431453/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT04431453/SAP_001.pdf